CLINICAL TRIAL: NCT03219099
Title: Population-Based Normative Database for HR-pQCT-Based Distal Radius and Tibia Strength Assessment in Switzerland
Brief Title: Normative Database for HR-pQCT-Based Radius and Tibia Strength
Acronym: NODARATIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: UKO-2017-1
Record Dates: First submitted 2017-07-13; First posted 2017-07-17 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Osteoporosis; Diagnoses Disease; Fracture; Bone Strength
MeSH Terms: conditions — Osteoporosis; Fractures, Bone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A novel methodology was recently developed and validated by the applicants to compute bone strength at the distal radius and tibia using second-generation HR-pQCT reconstructions. The methodology is expected to improve significantly the assessment of bone fracture risk in idiopathic and secondary osteoporosis, but no reference data and no reproducibility data are available.

The objective of the study is the determination of the sex- and age-specific distributions of accurate distal radius and tibia strength assessed by HR-pQCT in the Swiss population.

DETAILED DESCRIPTION:
Objective: De novo determination of sex- and age-specific reference intervals for vBMD, bone architecture, and bone strength assessed by 3D HR-pQCT with a resolution of 61 µm (Xtreme CT II, Scanco Medical, Brütisellen, Switzerland) in the Swiss population.

Design: Population-based, age- and sex-stratified, cross-sectional study in a single centre.

Study Size: For the main part, 480 valid data sets will be needed for two age reference intervals for both women and men. The number of double/triple stack scans will be between 1 and 3 depending on graded motion artefacts.

Among the 120 participants of each reference interval, 21 will be needed to assess reproducibility. For these volunteers, the number of double/triple stack scans will be equal to 3.

Project Assessments, Procedures: participant demographics and physical activity will be obtained and the validated Swiss FRAX questionnaire will be filled to determine the epidemiology-based 10-year fracture risk. Grip strength will be measured. A DXA measurement at the hip will be done according to the standard protocol of the Universitätspoliklinik für Osteoporose. For participants at elevated vertebral fracture risk, lateral and antero-posterior DXA of the spine will be added for vertebral fracture assessment (VFA) and spine areal bone mineral density (aBMD). The HR-pQCT examination per se consists then of up to 3 repeated double stack scans at the distal radius and triple stack scans at the distal tibia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged 20 years or older living in Switzerland
* Written informed consent

Exclusion Criteria:

* Psychological disorder or dementia in order to understand the informed consent and be able to fill the FRAX questionnaire
* Implant or a fracture at the DXA and HR-pQCT measurement sites
* Inability to keep the extremities still for the few minutes of an HR-pQCT examination (e.g. Parkinson disease or spastic syndrome)
* History of low trauma fracture
* Known pregnancy or lactating women
* History of hysterectomy and/or ovariectomy
* Known metabolic bone disorders, such as osteogenesis imperfecta, Paget's disease or sclerosteosis (osteopenia or idiopathic osteoporosis are not exclusion criteria)
* Ever use of one or more of the following bone active substances: bisphosphonates, RANKL-inhibitors (DENOSUMAB), selective estrogen receptors (SERMS) or parathormone/teriparatide
* Ever use of oral glucocorticoids during more than 3 months or currently taking glucocorticoids

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The project population are female and male healthy volunteers above 20 years old. Following international recommendations, the number of participants for the calculation of the reference intervals is set to 576. Among these, the assessment of reproducibility of the novel bone strength estimation methodology will be performed in 42 participants.
Sampling Method: Non-Probability Sample
Enrollment: 576 (Estimated)
Dates: Start 2018-06-14 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Bone strength at distal radius and tibia, assessed by HR-pQCT | At baseline (cross-sectional, single timepoint for data collection)
  Normative Database for HR-pQCT-Based Distal Radius and Tibia Strength in Swiss women and men

SECONDARY OUTCOMES:
In-vivo reproducibility of radius strength calculations | At baseline
  3 repeated double/ triple stack scans, after reposition, data collection within 1 hour at one single time point
In-vivo reproducibility of tibia strength calculations | At baseline
  3 repeated double/ triple stack scans, after reposition, data collection within 1 hour at one single time point

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Lippuner, M.D., Study Director — Department of Osteoporosis, Bern University Hospital, University of Bern, CH-3010 Bern, Switzerland; Philippe Zysset, Ph.D., Study Director — Institute of Surgical Technology and Biomechanics
Locations (1):
- University Hospital Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No